CLINICAL TRIAL: NCT00539942
Title: Extended Deep Venous Thrombosis Prophylaxis in Gynecologic Oncology Surgery With Intermittent Compression Devices (ICD) With or Without Postoperative Arixtra (Fondaparinux Sodium): A Randomized Controlled Trial
Brief Title: Study of Arixtra (Fondaparinux Sodium) to Prevent Blood Clots in Women Undergoing Abdominopelvic Surgery for Likely Gynecologic Malignancy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Problems with accrual
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Warner Huh, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F070727009; UAB 0723
Record Dates: First submitted 2007-10-03; First posted 2007-10-05 (Estimated); Results first posted 2012-03-09 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Venous Thrombosis
Keywords: Randomized Clinical Trials; Randomized Controlled Trial; Venous thrombosis; Anticoagulant Drugs; Doppler Ultrasound; Postoperative complications
MeSH Terms: conditions — Venous Thrombosis; Postoperative Complications | interventions — Fondaparinux; Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intermittent compression devices (ICD) (Active Comparator): All patients will receive intermittent compression devices (ICD's) during the patient's entire hospitalization after the operative procedure. Patients randomized to the standard of care management will receive ICD's only. This represents the current standard of care at our institution at the time of initiation of the trial.
  Interventions: Device: Intermittent compression devices (ICD)
- Arixtra (fondaparinux sodium) (Experimental): Patients randomized to treatment arm will initiate Arixtra (fondaparinux sodium) treatment on post-operative day 1 and continue treatment until post-operative day 22 (21 consecutive days). Subjects randomized to this arm are to receive the standard prophylactic dose for major abdominal surgery of 2.5 mg/day for a total of 21 consecutive days (including hospitalization time and after hospital discharge).
  Interventions: Drug: Arixtra (fondaparinux sodium)

INTERVENTIONS:
Drug: Arixtra (fondaparinux sodium) — Treatment will consist of daily injections of pharmacy prepared syringes of Arixtra (fondaparinux sodium) 2.5mg. Treatment will continue for 21 consecutive days to end on post-operative day 22.
  Arms: Arixtra (fondaparinux sodium)
Device: Intermittent compression devices (ICD) — All patients will receive intermittent compression devices (ICD's) during the patient's entire hospitalization after the operative procedure. Patients randomized to the standard of care management will receive ICD's only. This represents the current standard of care at our institution at the time of initiation of the trial.
  Arms: Intermittent compression devices (ICD)

SUMMARY:
This is a randomized trial to compare intermittent compression devices with or without post-operative Arixtra (fondaparinux sodium) in women undergoing major abdominal surgery for known or presumed gynecologic malignancies. This trial seeks to determine if there is a difference in the rate of deep venous thrombosis between these two groups.

DETAILED DESCRIPTION:
To assess the effectiveness of Arixtra (fondaparinux sodium) in the prophylaxis of deep venous thromboembolism in gynecologic oncology patients undergoing abdominopelvic surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing open laparotomy (non-laparoscopic) gynecologic surgery.
* Patients must be competent to self-administer injections, or must have caregivers or nurses who can perform injections
* Patients must have signed an approved informed consent

Exclusion Criteria:

* Patients with medical history which requires chronic anticoagulation (i.e. previous DVT, pulmonary embolism, atrial fibrillation, heart valve replacement)
* Patients with contraindications to anticoagulation (generalized bleeding disorders, peptic ulcer disease, hemorrhagic stroke, etc)
* Contraindications to placement of ICDs (history of lower extremity venous stasis ulcers)
* Patients receiving low molecular weight heparin or unfractionated heparin for prophylaxis post-operatively
* Patients who are unable to receive injections as an outpatient and/or unable to undergo a doppler ultrasound of the lower extremities
* Renal insufficiency (creatinine clearance < 30 mL/min)
* Patients who have a body weight < 50 kg
* Hypersensitivity to low molecular weight heparin
* Patients who are pregnant or have a positive pregnancy test.
* Patients receiving continuous (indwelling) epidural.

Ages: 19 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warner K. Huh, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Women's and Infant Center, 1700 6th Avenue South, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the UAB Gynecologic Oncology Practice from 4/2007 to 6/2010
Pre-assignment Details: Difficulty with recruiting subjects to this trial (subjects were not interested in participating)
Groups:
- Intermittent Compression Devices: Patients will receive standard intermittent compression devices (ICD's) during entire hospitalization after the operative procedure. Patients randomized to the standard of care management will receive ICD's only. This represents the current standard of care at our institution at the time of initiation of the trial.
- Arixtra (Fondaparinux Sodium): Patients randomized to treatment arm will initiate ARIXTRA treatment on post-operative day 1 and continue treatment until post-operative day 22 (21 consecutive days). Subjects randomized to this arm are to receive the standard prophylactic dose for major abdominal surgery of 2.5mg/day for a total of 21 consecutive days (this includes both while in the hospital and after hospital discharge)
Period: Overall Study
Arm/Group | Intermittent Compression Devices | Arixtra (Fondaparinux Sodium)
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fondaparinux (Arixtra): Patients randomized to treatment arm will initiate ARIXTRA treatment on post-operative day 1 and continue treatment until post-operative day 22 (21 consecutive days). Subjects randomized to this arm are to receive the standard prophylactic dose for major abdominal surgery of 2.5mg/day for a total of 21 consecutive days (this includes both while in the hospital and after hospital discharge)
- Total: Total of all reporting groups
Arm/Group | Intermittent Compression Devices | Fondaparinux (Arixtra) | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (12) | 57 (7) | 54 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Deep Venous Thromboembolism (DVT) Using Intermittent Compression Devices With and Without Arixtra
Description: Deep venous thromboembolism (DVT) rates are determined from lower extremity doppler ultrasound measurements.
Time Frame: 21 days
Population: Planned Intention to Treat analysis but was unable to complete due to inadequate number of subjects enrolled.
Measure: Number; unit: participants
Groups:
- Intermittent Compression Devices: Patients will receive intermittent compression devices (ICD's) during the entire hospitalization after the operative procedure. Patients randomized to the standard of care management will receive ICD's only. This represents the current standard of care at our institution at the time of initiation of the trial.
- Arixtra (Fondaparinux Sodium): Patients randomized to the Arixtra arm will initiate treatment on post-operative day 1 and continue treatment until post-operative day 22 (21 consecutive days). Subjects randomized to this arm are to receive the standard prophylactic dose for major abdominal surgery of 2.5 mg/day for a total of 21 consecutive days (including hospitalization and after hospital discharge)
Arm/Group | Intermittent Compression Devices | Arixtra (Fondaparinux Sodium)
Number analyzed (Participants) | 4 | 3
participants | 4 | 3
Statistical Analysis 1: Comparison: Intermittent Compression Devices vs Arixtra (Fondaparinux Sodium); Unable to analyze data; Test type: Superiority or Other; p < .05, Chi-squared; Mean Difference (Final Values) = 10

2. Secondary Outcome: Incidence of Untoward Effects With Arixtra
Description: Adverse events will be evaluated to determine untoward effects.
Time Frame: 21 days
Population: Unable to analyze data.
Measure: Number; unit: participants
Arm/Group | Intermittent Compression Devices | Arixtra (Fondaparinux Sodium)
Number analyzed (Participants) | 4 | 3
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Intermittent Compression Devices | Arixtra (Fondaparinux Sodium)
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/4 | 1/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermittent Compression Devices (N=4) | Arixtra (Fondaparinux Sodium) (N=3)
Pelvic Abscess (Reproductive system and breast disorders) | 1 (1) | 0 (0) — subject developed a pelvic abscess following a hysterectomy for leiomyomas
Postoperative Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) — subject developed a post-operative ileus following her surgery
Postoperative Death (Surgical and medical procedures) | 1 (1) | 0 (0) — subject expired at an outside hospital approximately month following surgery
Wound infection (Infections and infestations) | 0 (0) | 1 (1) — subject developed a wound infection following her surgery

LIMITATIONS AND CAVEATS:
This trial was terminated early due to poor enrollment and recruitment and the very small number of subjects analyzed. As such, the data is uninterpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less